CLINICAL TRIAL: NCT01368445
Title: Randomized, Double-Blind, Placebo-Controlled Trial of the Safety and Efficacy of MP03-36 in Patients With Seasonal Allergic Rhinitis
Brief Title: A Study to Evaluate the Safety and Efficacy of a Nasal Spray to Treat Seasonal Allergies
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Meda Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: MP433
Record Dates: First submitted 2011-06-06; First posted 2011-06-08 (Estimated); Last update posted 2011-10-06 (Estimated); Status verified 2011-10

CONDITIONS: Seasonal Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal | interventions — azelastine; Nasal Sprays

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- MP03-36 Nasal Spray (Active Comparator): azelastine hydrochloride 0.15%
  Interventions: Drug: azelastine hydrochloride 0.15% Nasal Spray
- MP03-36 and Placebo Nasal Spray (Active Comparator): azelastine hydrochloride 0.15% and Placebo
  Interventions: Drug: azelastine hydrochloride 0.15% and Placebo
- Azelastine 0.1%, Nasal Spray (Active Comparator): Azelastine 0.1%, Nasal Spray
  Interventions: Drug: Azelastine 0.1%, Nasal Spray
- Placebo Nasal Sapray (Placebo Comparator): 0mg, 2 sprays per nostril twice daily AM & PM)
  Interventions: Drug: azelastine hydrochloride 0.15% Nasal Spray; Drug: azelastine hydrochloride 0.15% and Placebo; Drug: Azelastine 0.1%, Nasal Spray

INTERVENTIONS:
Drug: azelastine hydrochloride 0.15% Nasal Spray — 1644 mcg, 2 sprays per nostril twice daily AM & PM)
  Other Names: astepro .15%
  Arms: MP03-36 Nasal Spray; Placebo Nasal Sapray
Drug: azelastine hydrochloride 0.15% and Placebo — 822 mcg azelastine hydrochloride 0.15%, 2 sprays per nostril once daily (AM) and 0mg placebo spray 2 sprays per nostril once daily (PM)
  Other Names: Astepro.15%
  Arms: MP03-36 and Placebo Nasal Spray; Placebo Nasal Sapray
Drug: Azelastine 0.1%, Nasal Spray — 1096 mcg, Azelastine 0.1%,2 sprays per nostril twice daily (AM & PM)
  Other Names: Astepro
  Arms: Azelastine 0.1%, Nasal Spray; Placebo Nasal Sapray

SUMMARY:
The Purpose of this study is to evaluate the safety and efficacy of MP03-36 (0.15% azelastine hydrochloride)at dosages of 2 sprays per nostril once daily and 2 sprays per nostril twice daily in patients with seasonal allergic rhinitis.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients 12 years of age and older
* Provide written informed consent/pediatric assent. If the patient is a minor, a parent or legal guardian must give written informed consent
* Screening Visit: Have a 12-hour reflective total nasal symptoms score ( TNSS) of at least 8 out of a possible 12 and a congestion score of 2 or 3 on Day -7
* Randomization Visit: Have a 12-hour reflective total nasal symptoms score (TNSS) (AM or PM) of at least 8 on 3 separate assessments (one of which was within 2 days of Day 1, and can include the morning of Day 1) during the Lead-in Period. In addition, an AM or PM nasal congestion score of 2 or 3 must have been recorded on 3 separate assessments (one of which was within 2 days of Day 1, and can include the morning of Day 1).
* Must have taken at least 10 doses of study medication during the lead-in period
* Randomization Visit: An instantaneous (TNSS) of ≥ 8 before beginning the onset of action assessment on Day 1
* Willing and able to comply with the study requirements
* At least a 2-year history of seasonal allergic rhinitis (SAR) during the fall pollen allergy season
* The presence of IgE-mediated hypersensitivity to local fall pollen confirmed by a positive response to either skin prick or intradermal testing within the last year. A positive response is defined as a wheal diameter of at least 3 mm larger than the control for the skin prick test or at least 7 mm larger than the control for the intradermal test.
* General good health and free of any disease or concomitant treatment that could interfere with the interpretation of the study results as determined by the investigator or the sponsor's medical officer
* Patients receiving immunotherapy injections (antigen desensitization) must be on a stable maintenance regimen for at least 30 days before the first study visit (adjustments to regimen following a brief period of missed injections does not preclude participation). Patients who are on maintenance doses of sublingual immunotherapy may be considered for the trial on a case-by-case basis after discussion with the sponsor's medical monitor or designee.

Exclusion Criteria:

* The use of any investigational drug within 30 days prior to Day -7. No investigational products are permitted for use during the conduct of this study
* Presence of any hypersensitivity to drugs similar to azelastine and to either sorbitol or sucralose (Splenda® brand sweetener)
* Women who are pregnant or nursing
* Women of childbearing potential who are not abstinent and not practicing a medically acceptable method of contraception
* Respiratory tract infections within two weeks prior to Day -7
* Respiratory Infections requiring oral antibiotic treatment two weeks prior to Day -7
* Other nasal disease(s) likely to affect deposition of intranasal medication, such as sinusitis, rhinitis medicamentosa or clinically significant polyposis or nasal structural abnormalities
* Patients with asthma (with the exception of mild, intermittent asthma)
* Patients with significant pulmonary disease
* Patients with a known history of alcohol or drug abuse
* Existence of any surgical or medical condition, which in the opinion of the investigator or sponsor, might significantly alter the absorption, distribution, metabolism, or excretion of study drug
* Clinically relevant abnormal physical findings within 1 week of randomization which, in the opinion of the investigator, would interfere with the objectives of the study or that may preclude compliance with the study procedures
* Planned travel outside the study area during the study period
* Family members and employees should be excluded
* Patients who received prohibited medications within specified timepoints in the protocol.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 617 (Actual)
Dates: Start 2006-08; Primary Completion 2006-11 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline in 12-hour reflective total nasal symptoms score(TNSS) for the entire 14-day study period compared to placebo | 14 Days

SECONDARY OUTCOMES:
Change from baseline in instantaneous total nasal symptoms score (TNSS) for the entire 14-day study period compared to placebo | 14 Days
Change from baseline to Day 14 in Roland Quality of Life Questionnaire (RQLQ )compared to placebo | 14 Days
Change From Baseline on Direct Visual Nasal Exams | 14 Days

CONTACTS AND LOCATIONS:
Locations (30):
- United States (30):
  - AABI Associates Medical Group, Fountain Valley, California
  - West Coast Clinical Trials, Long Beach, California
  - Allergy Research Foundation, Los Angeles, California
  - Southern California Research, Mission Viejo, California
  - Allergy Medical Group, Roseville, California
  - Allergy Associates Medical Group, San Diego, California
  - Allergy and Asthma Associates of CA, San Jose, California
  - The William Storms Allergy Clinic, Colorado Springs, Colorado
  - Colorado Allergy and Asthma Centers, PC, Denver, Colorado
  - Coastal Allergy and Asthma P.C., Savannah, Georgia
  - Kansas City Allergy and Asthma, Overland Park, Kansas
  - Institute for Asthma and Allergy, P.C., Wheaton, Maryland
  - Northeast Medical Research Associates, Inc., North Dartmouth, Massachusetts
  - Clinical Research Institute, Minneapolis, Minnesota
  - The Asthma and Allergy Center, PC, Papillion, Nebraska
  - Atlantic Allergy, Asthma & Immunology, Ocean City, New Jersey
  - Princeton Center for Clinical Research, Skillman, New Jersey
  - Allergy and Asthma Institue of Rochester, Rochester, New York
  - North Carolina Clinical Research, Raleigh, North Carolina
  - Clinical Research Center, Cincinnati, Ohio
  - Oklahoma Institute of Allergy and Asthma, Edmond, Oklahoma
  - Allergy and Asthma Consultants of NJ-PA, P.C, Collegeville, Pennsylvania
  - Valley Clinical Research Center, Easton, Pennsylvania
  - Allergy and Clinical Immunology Associates, Pittsburgh, Pennsylvania
  - Allergy Asthma Associates Research Dept., Austin, Texas
  - AARA Research Center, Dallas, Texas
  - Research Across America, Dallas, Texas
  - Central Texas Health Research, New Braunfels, Texas
  - Sylvana Research Associates, San Antonio, Texas
  - Allergy and Asthma Center, Waco, Texas